CLINICAL TRIAL: NCT02215148
Title: Pharmacokinetics and Clinical Response of Tolvaptan in Neurocritical Care Patients
Status: Terminated | Type: Observational
Why Stopped: Slow subject enrollment and contracting issues; sponsor decided to abort study
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Otsuka America Pharmaceutical (Industry); Medical University of South Carolina (Other); Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13-3991; 20141663 (Other Grant/Funding Number: Otsuka America Pharmaceutical, Inc.)
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Brain Injury; Hyponatremia
MeSH Terms: conditions — Brain Injuries; Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for pharmacokinetic sampling will be collected in serum separator tubes at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30 and 36 hours after the dose of study drug is administered. Serum sodium will be collected at baseline and 2, 4, 6, 8, 12, 24, and 36 hours after study drug administration. Approximately 180 mL of blood will be collected over 36 hours. Urinary output and urine specific gravity will be collected 0-2, 2-4, 3-6, 6-8, 8-12, and 12-24 hours after tolvaptan administration.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Brain injured patients with hyponatremia: Patients with acute brain injury who develop hyponatremia and are administered tolvaptan via the nasogastric tube, deemed necessary by the primary medical team.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan

SUMMARY:
To assess the pharmacokinetic profile of tolvaptan in critically ill acute brain injury patients and to secondarily evaluate the clinical response and safety of tolvaptan in acute brain injured patients

ELIGIBILITY:
Inclusion Criteria:

1. Acute brain injury patients in the ICU with hyponatremia (Na < 135 mmol/L) necessitating treatment in addition to fluid restriction per clinical judgement or patients at risk for worsening cerebral edema
2. Informed consent obtained from patient or authorized legal representative
3. Age ≥ 18 years

Exclusion Criteria:

1. Use of CYP3A4 inhibitors or inducers as medications, juices, or herbal supplements within 96 hours prior to the study period.
2. A positive urine or serum pregnancy test, or are currently breast-feeding
3. Patients with subarachnoid hemorrhage or in patients suspected to have cerebral salt wasting or any signs of volume depletion
4. Imminent death or brain death
5. Concomitant fungal infection
6. History of HIV
7. Concomitant administration of continuous infusion hypertonic saline, conivaptan or hypertonic saline bolus within 24 hours of study drug administration
8. Diuretic or mannitol administration within 6 hours
9. Serum creatinine ≥ 3.5 mg/dL
10. Diagnosis of cirrhosis or liver function tests > 2x the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be comprised of 30 acute brain injury patients in the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) and time to maximum observed plasma concentration (Tmax) of tolvaptan over 36 hours post-dose | Over 36 hours from drug administration
  Cmax will be derived from plasma concentrations versus time using a validated LS/MS/MS assay is sodium heparinized plasma. The tolvaptan assay has a range of 1.00 - 200 mg/mL. Blood samples will be collected at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30 and 36 hours after the dose of tolvaptan is administered. The first 15 patients will receive single dose 15mg of tolvaptan via a gastric tube and if determined not bioequivalent and no clinical response to oral administration and safe to administer, then last 15 patients will receive 30mg single dose via a gastric tube.
The elimination rate constant (ke) of tolvaptan over 36 hours post-dose | Over 36 hours from drug administration
  Ke derived from plasma concentrations versus time using a validated LS/MS/MS assay is sodium heparinized plasma. The tolvaptan assay has a range of 1.00 - 200 mg/mL. Blood samples will be collected at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30 and 36 hours after the dose of tolvaptan is administered. The first 15 patients will receive single dose 15mg of tolvaptan via a gastric tube and if determined not bioequivalent and no clinical response to oral administration and safe to administer, then last 15 patients will receive 30mg single dose via a gastric tube.
Area under the plasma concentration time curve (AUC) of tolvaptan from time zero to 36 hours post-dose | Over 36 hours from drug administration
  AUC will be computed from 0 to 36 hours using the linear-log trapezoidal method and extrapolated to infinity. Tolvaptan concentrations will be determined using a validated LS/MS/MS assay is sodium heparinized plasma. The tolvaptan assay has a range of 1.00 - 200 mg/mL. Blood samples will be collected at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30 and 36 hours after the dose of tolvaptan is administered. The first 15 patients will receive single dose 15mg of tolvaptan via a gastric tube and if determined not bioequivalent and no clinical response to oral administration and safe to administer, then last 15 patients will receive 30mg single dose via a gastric tube.

SECONDARY OUTCOMES:
The clinical response of tolvaptan administered through the nasogastric tube in acute brain injured patients | Over 36 hours from drug administration
  Clinical response is defined as a change in serum sodium of 4 - 6 mEq/L
The safety of tolvaptan administered via a nasogastric tube in acute brain injured patients | Over 36 hours from drug administration
  Safety assessments will include: vital signs, clinical laboratory tests, concomitant medications, and reported or observed adverse events. The rate of sodium correction will also be assessed. Excessive correction in sodium is defined as ≥ 12 mE/L increased in serum sodium within 24 hours of the dose. Excessive drop in blood pressure will be defined as >20% reduction in MAP from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Morbitzer, PharmD, Principal Investigator — University of North Carolina, Chapel Hill; Denise H. Rhoney, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina